CLINICAL TRIAL: NCT03376451
Title: Validation of Specific Biomarkers for the Diagnosis of Endometriosis
Brief Title: EndoSearch : Endometriosis Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Afchine Fazel (Industry)
Responsible Party: Sponsor-Investigator, Dr Afchine Fazel, MD PhD, Endodiag
Organization: Endodiag (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A01445-48
Record Dates: First submitted 2017-11-29; First posted 2017-12-18 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Endometriosis (Diagnosis); Blood Biomarkers; Endometrium Biomarkers
MeSH Terms: conditions — Endometriosis; Disease

STUDY DESIGN:
Intervention Model Description: EndoSearch recruits two groups of patients : affected by endometriosis and unaffected (controls) but both of them need a surgery for different indication (endometriosis for patients and other for controls (i.e dermoid cyst).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients in EndoSearch (Other): EndoSearch will conduct on only one cohort divided in two groups : patients affected by endometriosis and patient unaffected (controls). All of these patients need a laparoscopic surgery for endometriosis indication (endometriosis group) or another indication which is not endometriosis (controls). However, nothing in the surgery or the patient medical care will be different between the two groups : patients will be treated exactly the same.
  Interventions: Other: Assessment of endometrium and blood biomarkers for endometriosis diagnosis

INTERVENTIONS:
Other: Assessment of endometrium and blood biomarkers for endometriosis diagnosis — Biological samples will be collected from patients, sent to Endodiag, Paris, in France and be processed through IHC and molecular biology techniques to assess the ability of the identified biomarkers signature to diagnose and prognose endometriosis.

SUMMARY:
EndoSearch aims to analytically validate a cluster of specific biomarkers for endometriosis diagnosis and disease recurrence. This signature will be tested on endometrium and blood from 975 patients, divided in two groups : 550 patients affected by endometriosis and 225 patients unaffected (controls).

EndoSearch is not about drug or medical device assessment but a research study for biomarker analytical validation purpose.

DETAILED DESCRIPTION:
Endometriosis is a very common gynecological disease affecting 10% of women of reproductive age. Main symptoms are chronic and severe pain in pelvis area and infertility in up to 40% of affected women. Currently, the only method to obtain a reliable diagnosis is the analysis of endometriotic lesions removed during surgery under general anaesthesia. There is a real need to diagnosis endometriosis non-invasively and quickly in order to improve patient management.

EndoSearch aims to analytically validate a cluster of endometrial and blood biomarkers identified in previous studies and specific for the endometriosis diagnosis and disease prognosis recurrence. During 2 years (follow up period) and 9 months (inclusion period), 15 clinical centers worldwide will recruit patients and collect biological samples and personal and clinical data from these patients. The biological samples will be processed at Endodiag labs, Paris, France though lab biotechnology techniques. Results will allow the assessment of sensibility and specificity (NPV and PPV) of the biomarker signature for endometriosis diagnosis and disease recurrence.

ELIGIBILITY:
Inclusion Criteria for endometriosis patients :

* Woman, from 18 to 45
* Patients with endometriosis suspicion, associated adenomyosis is accepted
* Freely signature of the consent form
* Patient needs laparoscopy for endometriosis purpose (first intervention or recurrence) regardless of the endometriosis type (superficial, ovarian or deep)
* Possibility of follow up during 2 years.

Inclusion Criteria for Healthy voluntary patients:

* Woman 18 to 45
* Freely signature of the consent form
* Patient needs laparoscopy for another indication than endometriosis, adenomyosis, uterine fibroma & other fibroid pathologies (ex of surgeries: tubular sterilization, ovarian non-fibroid cyst, urinary incontinence requiring ureteral intervention).

Exclusion Criteria for endometriosis patients :

* Refusal or linguistic or psychic incapacity to sign informed consent
* No internet access or refusal to use new technologies
* Minor woman (under 18 years old)
* Pregnancy or breastfeeding
* Menopause
* Evidence of adenomyosis without endometriosis
* All metabolic pathology, endocrine, chronical infectious or malignant.
* Endometriosis negative result at visual and histological examination by anatomopathologist of the clinical centre.

Exclusion Criteria for Healthy voluntary patients

* Refusal or linguistic or psychic incapacity to sign informed consent
* No internet access or refusal to use new technologies
* Minor woman (under 18 years old)
* Pregnancy or breastfeeding
* Menopause
* Adenomyosis
* All metabolic pathology, endocrine, chronical infectious or malignant.
* Endometriosis positive result at visual and histological examination by anatomopathologist of the clinical centre.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Endometriosis is a gynecological disease so we are only recruiting female subjects.
Enrollment: 975 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensibility for endometriosis diagnosis (probability of detection) | Comparison between diagnosis lab result and anatomopathologist diagnosis at the end of inclusion phase (9 months after 1st patient inclusion)
  Measurement of the proportion of positives patient that are correctly identified as such for the endometriosis diagnosis.
Specificity for endometriosis diagnosis | Comparison between diagnosis lab result and anatomopathologist diagnosis at the end of inclusion phase (9 months after 1st patient inclusion)
  Measurement of the proportion of negatives patient that are correctly identified as such for the endometriosis diagnosis

SECONDARY OUTCOMES:
Sensibility for endometriosis recurrence prognostic (probability of detection) | Comparison between recurrence lab result and eCRF data on recurrence at the end of study (2 years and 9 months)
  Measurement of the proportion of positives patient that are correctly identified as such for the endometriosis recurrence prognostic.
Specificity for endometriosis recurrence prognostic | Comparison between recurrence lab result and eCRF data on recurrence at the end of study (2 years and 9 months)
  Measurement of the proportion of negatives patient that are correctly identified as such for the endometriosis recurrence prognostic.

CONTACTS AND LOCATIONS:
Locations (1):
- Endodiag, Paris, France

IPD SHARING:
Plan to Share IPD: No